CLINICAL TRIAL: NCT03731156
Title: Biological Diagnosis of Granulomatous Pneumocystis Pneumonia
Brief Title: Granulomatous Pneumocystis Pneumonia
Acronym: NC
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0422
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Pulmonary Nodule; Invasive Fungal Infections; Pneumocystis Jirovecii
Keywords: Granulomatous Pneumocystis Pneumonia; PCR Pneumocystis jirovecii
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The intra-alveolar form of Pneumocystis jiroveci pneumonia (PjP) is a common pathology in immunocompromised patients, particularly those infected with HIV. The diagnosis is based on the detection of Pj in a LBA. Intra-tissue granulomatous form (PGP) is a rare entity observed in non-HIV immunocompromised patients. In this case, the LBA is mostly non-contributory and the diagnosis is based solely on the detection of cysts on histological examination on biopsy of a pulmonary nodule. For many years, it has been clearly demonstrated that the use of a specific PCR clearly improves the biological diagnosis of PcP. However, in case of granulomatous form this method is not implemented because the diagnostic hypothesis is not mentioned.

In 2018, two cases of PGP were diagnosed at 3-month intervals at Montpellier University Hospital Center. The diagnostic confirmation was obtained with PCR Pj. In this context the investigators will investigate the interest of implementing PCR Pj on biopsies on pulmonary nodules from hospitalized patients between 2015 and 2018. In all selected patients, histopathological aspect of the nodule was compatible with a PGP and, no other diagnosis has been confirmed (infectious, tumoral, inflammatory ...). Finally, 17 patients were selected to check retrospectively, if the presence of Pj could be at the origin of the pathology.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary nodule

Exclusion Criteria:

* nodule : tumoral, other infections than Pj, inflammatory

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodule
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
PCR results | 1 day
  PCR results

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Lachaud, MD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC